CLINICAL TRIAL: NCT04849429
Title: A Randomized, Double-blind Controlled Trial of the Efficacy of an Intra-discal Injection of Autologous Platelet-rich Plasma (PRP) Enriched With Exosomes (PRPex) Versus Placebo in Chronic Low Back Pain
Brief Title: Intra-discal Injection of Platelet-rich Plasma (PRP) Enriched With Exosomes in Chronic Low Back Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Himanshu Bansal Foundation (Other)
Responsible Party: Principal Investigator, anupama agrawal, Principal Investigator, Dr. Himanshu Bansal Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HB/CLINICALTRIAL/01/2021
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Chronic Low Back Pain; Degenerative Disc Disease
Keywords: intra-discal PRPEx Chronic Low Back Pain
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: 1. Arm I will be assigned to receive placebo (trigger point injection under carm)
  2. Arm II: to receive PRP with exosomes at the center of the nucleus pulposus (2ml)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be randomly selected based on computer generated number to receive one undistinguishable injection of PRP ex or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (trigger point injection under C-arm)
  Interventions: Drug: Normal Saline
- Platelet rich plasma (PRP) with exosomes (Experimental): PRP with exosomes at the center of the nucleus pulposus (2ml)
  Interventions: Biological: Platelet rich plasma (PRP) with exosomes

INTERVENTIONS:
Biological: Platelet rich plasma (PRP) with exosomes — Autologous Platelet rich plasma (PRP) with exosomes Following skin disinfection of the back 2 ml from the total PRPex procured will be injected as soon as possible by an fluoroscopy guided lateral approach.
  Arms: Platelet rich plasma (PRP) with exosomes
Drug: Normal Saline — placebo : 2 ml normal saline para discal administration
  Arms: Placebo

SUMMARY:
Intervertebral disc pathology accounts for 40% or more cases of chronic LBP. Available treatment options do not improve the underlying degenerative condition hence This indicates the need for new therapies.

intradiscal injection of PRP with exosomes derived from blood may potentially transmit some of the unique stem cell properties to other stem cells, facilitating stemness maintenance, differentiation, self-renewal, and repair.

controlled, randomized, double-blind placebo clinical trial to compare the safety and efficacy of PRP with exosomes in discogenic LBP adminstartion of PRP with exosomes at the centre of the nucleus pulposus or equal amount of placebo paradiscal patients wil be elvaluated for primary Outcome measures viz: Visual analog scale (VAS), Roland Morris Disability Questionnaire (RDQ), SF 36 health questionnaire, Functional rating index and Secondary: MRI - disc degeneration grading, T2 quantification, and for any Adverse events including of discitis

DETAILED DESCRIPTION:
Management of chronic low back pain (LBP) has contributed to its high socioeconomic The intervertebral disc accounts for 40% or more cases of chronic LBP. Available treatment options do not improve the underlying degenerative condition, although they do resolve its symptoms. This indicates the need for new therapies and/or interventions that actually treat the underlying causes of discogenic pain. Biological therapies by direct injection of PRP into the annulus fibrosus and nucleus pulposus seems an effective and feasible option.

Exosomes derived from blood may potentially transmit some of the unique stem cell properties to other stem cells, facilitating stemness maintenance, differentiation, self-renewal, and repair.

We propose to have a controlled, randomized, double-blind clinical trial to compare the safety and efficacy of exosomes in LBP. Informed consent will be obtained from all subjects prior to study participation.

PRP Preparation:

Blood sample (60 ml) will be centrifuged at 600×g for 10 min to collect plasma fraction. And centrifuged at 4000×g for 15 min. Supernatant platelet poor plasma (PPP) will be then removed, leaving 1 ml PRP. PPP will be passed through one-micron special indigenous designed flush back filter (Alpha Corpuscle, Delhi, India) so that all the platelets present in PPP fraction will get trapped in the filter. These trapped platelets will be flushed back with 1 ml of PPP to retrieve most of the platelets. This will be mixed together and then passed through a WBC filter (Terumo Imuguard, USA) to filter off the leukocytes. The final PRP concentrate (0.1 ml) will be analysed for total leukocyte & platelet counts. Five samples will be selected randomly treated with bovine thrombin reconstituted in 10% calcium chloride will be assessed for growth factors [platelet-derived growth factors (PDGF) and vascular endothelial growth factors (VEGF)] by ELISA.

On an average our PRP sample will have 100 billion platelets and 30x concentrate of blood platelet in 2ml of final PRP.

Exosomes preparation:

Sixty ml of blood in EDTA-coated tubes will be spin at 1,200 g for 10 minutes at 4°C to separate plasma. Plasma will be filtered with (0.22 μm) filter. Avoid any pelleted material while transferring the plasma. Discard the pelleted material. This tube has special filter to concentrate exosomes and other growth promoting proteins. Tube will be centrifuged at 3000 g, RT, 30 min and exosomes will be collected and then will be concentrated (0.5 ml to 3ml). To recover exosomes clogged in wall of filter -add 20 ml NS (preferably PBS) into micro centrifuge tube and rinsed it by centrifugation at 3,500 g. Collect the concentrated soup of exosomes again which were clogged in filter wall.

Quantification of protein content will be done by bicinchoninic acid (BCA) assay.

Nanoparticle tracking analysis (NTA) Vesicle suspensions with concentrations between 1×107/ml and 1×109/ml will be examined using a Nanosight NS300 (NanoSight Ltd., UK) equipped with a 405 nm laser to determine the size and quantity of particles isolated. A video of 60-sec duration will be taken with a frame rate of 30 frames/sec, and particle movement will be analyzed using NTA software (version 2.3; NanoSight Ltd.).

Western blot analysis The exosome supernatant will be denatured in sample buffer and will be subjected to western blot analysis. Purified exosomes will be analysed for protein expression HSP70, flottilin, CD63, TSG101 and calnexin. The proteins were visualized on the Bio-Rad ChemiDoc XRS Imager system (Bio-Rad Laboratories, Berkeley, CA, USA).

Study Design Patients will be randomized into 2 arms with either to receive PRP with exosomes at the centre of the nucleus pulposus or equal amount of placebo and will be evaluated by 2 interventional spine and medicine physicians.

Randomisation and Arms of the study:

Approximately Three hundred patients will be screened to randomly allocate to treatment or control groups at a 1:1 ratio, to assign 30 patients into each 4 arm:

1. Arm I will be assigned to receive placebo (trigger point injection under C arm)
2. Arm II: to receive PRP with exosomes at the center of the nucleus pulposus (2ml) Test product(s), dose and mode of administration duration of treatment Patients will be randomly selected based on computer generated number to receive one undistinguishable injection of PRP ex or placebo. Following skin disinfection of the back 2 ml from the total PRPex procured was injected as soon as possible by an fluoroscopy guided lateral approach. Patients received the placebo in a similar manner but not to disc .it will be in muscles zone around trigger point .Physician who evaluated the study and patient were unknown of treatment. Patients were advised to continue with usual exercises, routine precautions, physiotherapy and back care.

   Paracetamol (to a maximum of up to one gram) three times a day, will be allowed to be used as a rescue drug. No systemic corticosteroid, potential symptom-modifying drug /procedure will be allowed during the study.

   Study assessments / Outcome measures
   1. Visual analog scale (VAS)
   2. Roland Morris Disability Questionnaire (RDQ)
   3. SF 36 health questionnaire
   4. Functional rating index
   5. MRI - disc degeneration grading, T2 quantification any evidence of discitis Patients will be assessed by visual analog scale (VAS), SF 36 health questionnaire, Functional rating index at baseline and followed at 1, 3, 6, and 12 months. The structural efficacy will evaluated by MRI t2 quantification and grading as described earlier in literature at baseline and at 6 months by two experienced radiologists. Assessors will be blinded.

      Monitoring visits will be conducted according to standard monitoring procedures.

      Discontinuation from treatment with a specific reason will be ascertained. Any evidence of infection/discitis will be delicately observed. Worsening of pain will be deeply analyzed.

      The patients will be evaluated for any adverse effects and vital signs once a week for the first month and then once a month up to 6 months. Blood samples were collected at the time of entry into the study, at six months, and on a final visit to examine biological variables as well as liver and kidney functions. Tolerability was assessed and laboratory-based haematological and biochemical assays were performed. A possible causal relationship with the treatment arm will also be assessed.

      STATISTICAL ANALYSIS:

      Analysis of variance (ANOVA) will be used to investigate the differences between groups. Differences in paired samples will be compared using the two-tailed Student's t-test. Correlations between variables will be assessed by Pearson's correlation. SPSS 20.0 will be used for statistical analyses (SPSS, Inc., Chicago, IL, USA). P<0.05 will be considered to be statistically significant.

      Identification of the relationship between safety issues/side effects and arousal level using measurement by rating scales. To test whether the relationship between safety issues/side effects and arousal level differs between IBRF ACP/MCP vs. Standard of Care groups, using measurement by rating scales, two analyses will be conducted. Canonical correlation will be used to determine which side effect (or combination of side effects) explains variance in the rating scale measurements. Additionally, cluster analysis will be employed to determine whether side effects are similarly related to arousal levels and outcomes for patients in the three treatment groups.

      MONITORING PROCEDURES/ADVERSE EVENTS / SAFETY ENDPOINTS Monitoring The monitors will visit the center during the study in addition to maintaining frequent telephone and written communication.

      The following guidelines meet the requirements specified in 21 CFR §812.46 and are provided to describe the procedures for monitoring the clinical studies. If the investigator is not complying with the signed Investigator Agreement, the protocol, or any condition of the study (e.g., incomplete data forms), the monitor has the right to terminate the investigator's participation in the study.

      Pre-Study Monitoring Procedures

      The designate (i.e. monitor) will be responsible for determining and documenting that each investigator clearly understands and accepts the responsibilities and obligations incurred in conducting a clinical study. The monitor will ensure prior to study initiation that the investigator:

      • Understands the requirements for a well-controlled study;

      • Understands the nature of the clinical protocol

      • Understands his/her reporting obligations;

      • Understands the requirements for device accountability;

      • Understands and accepts the obligations to obtain informed consent in accordance with 21 CFR Parts 50 and 56;

      • Understands and accepts the obligation to obtain IRB review and approval of the clinical investigation before it is initiated and to ensure continuing review of the study by the IRB in accordance with 21 CFR Part 56, and to keep the sponsor informed of all IRB actions concerning the study;
      * Understands and accepts the requirements regarding financial disclosure of clinical investigations, 21 CFR Part 54;
      * Has adequate facilities and access to an adequate number of suitable subjects to conduct the investigation;
      * Has the required documentation on file, including IRB approval and a signed investigator agreement.

      Periodic Monitoring Visits • Monitoring visits will be conducted in accordance with the FDA Guideline for the Monitoring of Clinical Investigations - January 1988.

      • The monitor should visit each site regularly to ensure the following:

      • Facilities continue to be adequate and acceptable.

      • The protocol is being properly followed.

      • The IRB/IEC has approved or been notified of any protocol changes.

      • Accurate, complete and current records are being maintained, and the information recorded.

      • Accurate, complete and timely adverse event reports are being submitted

      • Informed consent has been obtained.

      • The reason for a subject's withdrawal from the study has been documented.

      • Reports are being submitted to the IRB and sponsor.

      • The appropriate staff is carrying out study activities.

      • All case report forms and other documentation related to the study will be reviewed upon receipt, and the site will be promptly notified of any deficiencies.

      Frequency of Monitoring Visits a) Monitoring visits will be conducted according to standard monitoring procedures. Monitoring visits will be determined on the basis of several factors, including: b) Duration of the study; c) Number of outstanding issues from previous visits; d) Number of subjects enrolled; e) Number of investigators/sites; and, f) Complexity of the study.

      Study Termination All routine monitoring functions must be performed prior to the study termination visit. The study termination visit may be combined with a monitoring visit. The following tasks should be completed at the last visit by the monitor.

   <!-- -->

   1. Remind the investigator of the obligation to retain the records. b) Prepare final monitoring report for IEC.

   Reports of Monitoring Visits

   Monitoring reports must be completed for all visits. Reports must include the following information:

   a) Date of the visit; b) List of study site personnel present; c) A summary of the findings, problems

ELIGIBILITY:
Inclusion Criteria:

1. Age between18 Years to 60 Years of any sex 2. Written and signed informed consent form 3. Chronic low back pain without leg pain for more than 3 months. 2. Symptomatic moderate to severe discogenic low back pain as defined according to the following criteria: centralized chronic low back that increased with activity and lasted at least six months.

3. Failure of conservative treatment measures (oral medications, rehabilitation therapy, and/or injection therapy) 4. Evidence of degeneration, as indicated via magnetic resonance imaging (MRI) decreased signal intensity on T2.

5. MRI Pfirrmann (MRI) score 3-6 6. Modic Grade II change or less 7. Disk protrusion less than 5 mm on magnetic resonance imaging maintenance of 50% or more of normal disc height. An intact annulus is not required 8. Subjects must be able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

1. Spinal stenosis
2. An abnormal neurologic exam
3. Symptomatic compressive pathology
4. A disc herniation causing significant compression with neurologic deficit.
5. Extrusions or sequestered disk fragments
6. Any spondylolisthesis or spondylolysis.
7. Presence of a grade 5 annular fissure on discography

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Change from Baseline VAS at 1,3, 6,12 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain. Change in VAS score will be assessed.
Roland Morris Disability Questionnaire (RDQ) | Change from Baseline RDQ at 1,3,6,12 months
  The Roland-Morris is a 24-item self-report questionnaire about how low-back pain affects functional activities. Each question is worth one point so scores can range from 0 (no disability) to 24 (severe disability)
SF 36 health questionnaire | Change from Baseline SF 36 at 1,3,6,12 months
  The SF.36 questionnaire (SF-36) contains 36 items that assess patients' health status and its impact on their lives. It comprises 36 questions which cover eight domains of health
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions. Change in SF 36 will be assessed.
Functional rating index | Change from Baseline Functional rating index at 1,3,6,12 months
  The Functional Rating Index (FRI) is an instrument specifically designed to quantitatively measure the subjective perception of function and pain of the spinal musculoskeletal system. Change will be assessed.

SECONDARY OUTCOMES:
MRI | Changes from baseline MRI findings will be assesed at 12 months
  magnetic resonance imaging to quantify grading of disc degeneration. *Grades 1, 2, and 3 are based on the signal intensity of the nucleus and inner fibers of anulus. For Grade 4, the margins between the inner and other fibers of the anulus at the posterior margin of the disc are indistinct.
  For Grade 5, the disc is uniformly hypointense, although there is no loss of disc space height. For Grades, 6, 7, and 8, there is progressive loss of disc space height. These could be broadly classified as mild, moderate, to severe loss of disc space height.
  Pfirrmann scoring Modic Grade

CONTACTS AND LOCATIONS:
Overall Officials: HIMANSHU BANSAL, MS, Principal Investigator — HIMANSHU BANSAL FOUNDATION; JEREMY PONT, Mchiro, Principal Investigator — PHOENIX HELSE Norway; DAVID WILSON, MBBS, Principal Investigator — PHOENIX HELSE Norway
Locations (2):
- India (2):
  - Anupam Hospital, Rudrapur, Uttarakhand
  - Mother Cell Spinal Injury and Stem Cell Research, Anupam Hospital, Rudrapur, Uttarakhand

IPD SHARING:
Plan to Share IPD: Yes
ANYTHING ASKED WILL BE SHARED ANYTIME
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: ANYTIME
Access Criteria: ANYONE INTERESTED TO CRITICALLY EVALUATE OR REPRODUCE
URL: http://DRHBF.ORG